CLINICAL TRIAL: NCT06103591
Title: Controlled Arterial Protection to Ultimately Remove Embolic Material
Acronym: CAPTURE-1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: EmStop Inc (Industry)
Collaborators: Bright Research Partners (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: EMS-CL-5000
Record Dates: First submitted 2023-10-19; First posted 2023-10-27 (Actual); Results first posted 2025-04-29 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Aortic Valve Stenosis
Keywords: Transcatheter Aortic Valve Replacement; Aortic Valve Replacement
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- EmStop Embolic Protection System (Experimental): Transcatheter aortic valve replacement (TAVR) procedures with the EmStop Embolic Protection System (EmStop System).
  Interventions: Device: The EmStop Embolic Protection System (EmStop System)

INTERVENTIONS:
Device: The EmStop Embolic Protection System (EmStop System) — The EmStop Embolic Protection System (EmStop System) is a catheter-based filter system that captures and removes debris dislodged during transcatheter aortic valve replacement (TAVR) procedures.

SUMMARY:
The objective of this study is to demonstrate device feasibility, safety and investigate performance of the EmStop Embolic Protection System when used as indicated in 15 subjects at 2 investigational sites in the U.S.

DETAILED DESCRIPTION:
The investigation is a prospective, multi-center, single arm feasibility study. Subjects will undergo treatment with a currently marketed TAVR device and the EmStop Embolic Protection System and will then be followed to 30 days post-procedure. This is a treatment-only feasibility investigation intended to capture and characterize outcomes, especially safety outcomes, with the EmStop System.

ELIGIBILITY:
Inclusion Criteria:

Clinical & Angiographic Inclusion Criteria

1. Between 21 and 90 years of age at the time of consent
2. Meets FDA approved indications for transcatheter aortic valve replacement (TAVR) procedure on a native aortic valve using a commercially available Abbott or Medtronic transcatheter heart valve
3. Willing and able to provide written informed consent and written HIPAA authorization prior to initiation of study procedures
4. Willing and able to comply with the protocol-specified procedures and assessments
5. Subject anatomy is compatible with correct device deployment and positioning with:

   * Ability to achieve access with a 21 French equivalent femoral access sheath
   * Ascending aorta length ≥8 cm
   * Ascending aorta/aortic arch diameter is ≥25 or ≤40 mm
   * Ascending aorta or aortic arch exhibits ≤ Grade 1 atheromatous disease and limited wall calcification

Exclusion Criteria:

1. Requires urgent or emergent TAVR procedure
2. Contraindicated to MRI
3. Previously implanted aortic or mitral valve bioprosthesis
4. Hepatic failure (Child-Pugh class C)
5. Hypercoagulable state that cannot be corrected by additional periprocedural heparin
6. Planned to undergo any other cardiac surgical or interventional procedure (e.g., concurrent coronary revascularization) during the TAVR procedure or within 30 days prior to the TAVR procedure. NOTE: Diagnostic cardiac catheterization is permitted up until baseline MRI is obtained. Once baseline MRI is obtained, no additional intra-aortic or intracardiac procedure may occur.
7. Acute myocardial infarction within 30 days of the planned index procedure
8. Renal failure, defined as estimated glomerular filtration rate (eGFR) <30 mL/min
9. Documented history of stroke or TIA within the prior 6 months, or any prior stroke with a permanent major disability or deficit (NIHSS >1 at baseline)
10. Left ventricular ejection fraction ≤30% within 3 months prior to procedure
11. History of intolerance, allergic reaction, or contraindication to any of the study medications, including heparin, aspirin, clopidogrel, or a sensitivity to contrast media or anesthesia that cannot be adequately pre-treated
12. Known allergy or sensitivity to nickel-titanium
13. Active endocarditis or ongoing systemic infection, defined as fever (>38°C) and/or white blood cell (WBC) >15,000 IU
14. Undergoing therapeutic thrombolysis
15. History of bleeding diathesis or a coagulopathy
16. Known or suspected to be pregnant, or is lactating; female subjects of child-bearing potential must have a negative serum or urine pregnancy test within 48 hours prior to the index study procedure.
17. Currently participating in another drug or device clinical study
18. Any other clinical reason, as deemed by the investigators of the study, by which the patient would not be an appropriate candidate for the study
19. Vulnerable subject populations (e.g., incarcerated or cognitively challenged adults)

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2023-12-27 (Actual); Primary Completion 2024-09-04 (Actual); Study Completion 2024-10-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emily Vollbrecht, Study Director — Bright Research Partners
Locations (2):
- United States (2):
  - Mission Health, Asheville, North Carolina
  - Centennial Medical Center, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | EmStop Embolic Protection System
Started | 15
Completed | 14
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | EmStop Embolic Protection System
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 79.07 (5.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 15
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Procedural Success
Description: Defined as successful insertion, deployment, positioning, and removal of the EmStop System in the absence of device interference
Time Frame: During the procedure
Measure: Count of Participants; unit: Participants
Arm/Group | EmStop Embolic Protection System
Number analyzed (Participants) | 15
Participants | 14

2. Primary Outcome: Occurrence of Major Adverse Cardiac and Cerebrovascular Events (MACCE) at 30 Days
Description: Defined as composite of the VARC-2 defined components (all-cause mortality, all stroke (disabling and non-disabling), acute kidney injury stage 2 or 3 (including renal replacement therapy) within 72 hours)
Time Frame: 30 days follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | EmStop Embolic Protection System
Number analyzed (Participants) | 15
Participants
  All-cause mortality | 1
  All stroke (disabling and non-disabling) | 1
  Acute kidney injury stage 2 or 3 (including renal replacement therapy) within 72 hours | 0

3. Secondary Outcome: Average Number of Captured Embolic Debris
Description: Device filters were shipped to an independent pathology core laboratory where debris were counted and assessed
Time Frame: During the procedure
Measure: Mean (Standard Deviation); unit: total number of captured particles
Arm/Group | EmStop Embolic Protection System
Number analyzed (Participants) | 15
total number of captured particles | 3169.00 (2059.30)

4. Secondary Outcome: Average Number of Captured Particles ≥140 μm in Diameter
Description: Assessed by an independent pathology core laboratory
Time Frame: Procedural
Measure: Mean (Standard Deviation); unit: total number of captured particles
Arm/Group | EmStop Embolic Protection System
Number analyzed (Participants) | 15
total number of captured particles | 3169.00 (2059.30)

5. Secondary Outcome: Total Acute Infarct Burden
Description: As measured by diffusion-weighted imaging (DWI), also referred to as DW-MRI. A baseline DW-MRI was collected and evaluated in comparison to the post-procedure DW-MRI.
Time Frame: 14 days pre-procedure to 18-36 hours post-procedure
Measure: Mean (Standard Deviation); unit: lesions
Arm/Group | EmStop Embolic Protection System
Number analyzed (Participants) | 15
lesions | 14.93 (12.62)

6. Secondary Outcome: Occurrence of Transient Ischemic Attack (TIA)
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | EmStop Embolic Protection System
Number analyzed (Participants) | 15
Participants | 0

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected from the time of subject enrollment through final 30 day follow-up and were adjudicated by an independent medical monitor.
Description: Adverse events were assessed at all visit timepoints (pre-discharge and 30-day follow up).
Arm/Group | EmStop Embolic Protection System
All-Cause Mortality (participants affected / at risk) | 1/15
Serious Adverse Events (participants affected / at risk) | 6/15
Other Adverse Events (participants affected / at risk) | 4/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EmStop Embolic Protection System (N=15)
1st Hb with Intermittent Complete Heart Block (Cardiac disorders) | 1 (1)
Stroke with metabolic encephalopathy and cardiac arrest (Cardiac disorders) | 1 (1)
Silent brain infarction (Nervous system disorders) | 1 (1)
Complete Heart Block (Cardiac disorders) | 1 (1)
Atrioventricular Block (Cardiac disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Symptomatic Bradycardia (Cardiac disorders) | 1 (1)
Decompensated Heart Failure (Cardiac disorders) | 1 (1)
SVT Involving the Cephalic Vein (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EmStop Embolic Protection System (N=15)
New Onset Left Bundle Branch Block; Nonspecific St Abnormality; Nonspecific Intraventricular Block (Investigations) | 1 (1)
Conduction System Injury (Cardiac disorders) | 1 (2)
Dizziness (Nervous system disorders) | 1 (1)
Virus (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-10-10): https://cdn.clinicaltrials.gov/large-docs/91/NCT06103591/Prot_SAP_000.pdf